CLINICAL TRIAL: NCT04637178
Title: Identifying Molecular Determinants for the Efficacy of Resistance Training for Improving Endurance Performance in Elite Cyclists
Brief Title: Predicting the Efficacy of Resistance Exercise Training for Improving Endurance Performance
Acronym: IDperform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trainome 2020#025-2
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-11

CONDITIONS: Elite Cyclists
Keywords: Cycling; Endurance performance; Skeletal muscle biology; Individualization; Muscle fiber type proportions; Ribosomal RNA
MeSH Terms: interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants/investigators will be blinded to muscle biological charateristics until after clean-up of main outcome variables. Participants/investigators will be aware of intervention arm affiliation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training added to endurance training (Experimental): Participants (elite cyclists) will conduct heavy-load resistance training twice a week in addition to their habitual endurance training for ten weeks
  Interventions: Behavioral: Resistance training; Behavioral: Endurance training (habitual)
- Endurance training (Other): Participants (elite cyclists) will conduct habitual endurance training-only for ten weeks
  Interventions: Behavioral: Endurance training (habitual)

INTERVENTIONS:
Behavioral: Resistance training — Resistance training sessions twice a week for ten weeks
  Other Names: Heavy-load strength training
  Arms: Resistance training added to endurance training
Behavioral: Endurance training (habitual) — Endurance training for ten weeks (habitual routines)

SUMMARY:
The overall objective of the study is to identify molecular determinants of the efficacy of resistance training for improving endruance performance in elite cyclists

DETAILED DESCRIPTION:
For elite endurance athletes, the addition of resistance training to habitual endurance training routines generally leads to improved endurance performance. However, this is not always the case, with several individuals failing to respond in the expected manner. This inter-individual variation is likely associated with inherent cellular and molecular charateristics of skeletal muscle. Indeed, responses to resistance training seem to be associated with muscle biological characteristics such as muscle fiber composition and ribosomal content (during the early phase of resistance training).

The study will investigate the association between muscle fibre composition (type I vs type II muscle fiber proportions) / ribosomal content in m. vastus lateralis and the effects of 10 weeks of resistance training on endurance performance in 52 elite cyclists. Half the participants will perform resistance training in addition to their habitual endurance training routines, the other half will perform endurance training-only. Muscle biopsies will be sampled from m. vastus lateralis before and after the first two weeks of the intervention. For muscle fiber composition, the hypothesis is that larger proportions of type II fibers will be associated with more pronounced benefits of resistance training. For ribosomal content, the hypothesis is that higher rRNA content at baseline and larger increases in rRNA content during the initial part of the intervention will be associated with more pronounced benefits of resistance training. No changes are expected in the non-resistance training control group.

ELIGIBILITY:
Inclusion criteria:

* VO2max > 65 ml/kg/min (male participants)
* VO2max > 50 ml/kg/min (female participants)
* >7 hours of endurance training per week for the 6 months leading up to the study

Exclusion criteria:

- having conducted regular resistance training for the last 6 months leading up to the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Performance during a 40-minute all-out cycling test | Changes from before the intervention to immediately after the intervention
  Mean power output measured during a 40-minute all-out cycling test
Performance during a 15-minute all-out cycling test | Changes from before the intervention to immediately after the intervention
  Mean power output measured during a 15-minute all-out cycling test

SECONDARY OUTCOMES:
Total RNA in muscle tissue (before intervention) | Before the intervention
  Total RNA content in m. vastus lateralis (ug per mg tissue)
Total RNA in muscle tissue (changes after two weeks) | Changes from before the intervention to immediately after the initial two weeks of resistance training
  Total RNA content in m. vastus lateralis (ug per mg tissue)
Muscle fiber proportions (before intervention) | Before the intervention
  Muscle fiber proportions in m. vastus lateralis measured using immunohistochemistry
Muscle fiber proportions (changes after two weeks) | Changes from before the intervention to immediately after the initial two weeks of resistance training
  Muscle fiber proportions in m. vastus lateralis measured using immunohistochemistry
Muscle fiber cross-sectional area (before intervention) | Before the intervention
  Cross-sectional area of muscle fibres in m. vastus lateralis measured using immunohistochemistry
Muscle fiber cross-sectional area (changes after two weeks) | Changes from before the intervention to immediately after the initial two weeks of resistance training
  Cross-sectional area of muscle fibres in m. vastus lateralis measured using immunohistochemistry
Myonuclear number (before intervention) | Before the intervention
  Myonuclei per muscle fiber in m. vastus lateralis measured using immunohistochemistry
Myonuclear number (changes after two weeks) | Changes from before the intervention to immediately after the initial two weeks of resistance training
  Myonuclei per muscle fiber in m. vastus lateralis measured using immunohistochemistry
rRNA expression (before intervention) | Before the intervention
  rRNA abundances in m. vastus lateralis measured using qPCR
rRNA expression (changes after two weeks) | Changes from before the intervention to immediately after the initial two weeks of resistance training
  rRNA abundances in m. vastus lateralis measured using qPCR
mRNA expression (before intervention) | Before the intervention
  mRNA abundances in m. vastus lateralis measured using qPCR
mRNA expression (changes after two weeks) | Changes from before the intervention to immediately after the initial two weeks of resistance training
  mRNA abundances in m. vastus lateralis measured using qPCR
Maximal concentric force production | Changes from before the intervention to immediately after the intervention
  Maximal concentric force production measured using a seated leg press test
Sprint performance | Changes from before the intervention to immediately after the intervention
  Mean power output measured during a 10-second all-out cycling sprint
Maximal oxygen consumption | Changes from before the intervention to immediately after the intervention
  Maximal oxygen consumption measured during an incremental cycling exercise test to exhaustion
Maximal aerobic power output | Changes from before the intervention to immediately after the intervention
  Maximal aerobic power output measured as mean power output during the last minute of an incremental cycling exercise test to exhaustion
Power output at lactate threshold | Changes from before the intervention to immediately after the intervention
  Power output at 4 mmol blood lactate concentration measured during an incremental cycling exercise test (with 5 minute steps)
Gross efficiency | Changes from before the intervention to immediately after the intervention
  Contribution of total energy turnover to power output in the fresh and fatigued state
Fractional utilization of VO2max (incremental test) | Changes from before the intervention to immediately after the intervention
  Fractional utilization of VO2max measured at 4 mmol blood lactate concentrations measured during an incremental cycling exercise test (with 5 minute steps)
Fractional utilization of VO2max (15-minute performance test) | Changes from before the intervention to immediately after the intervention
  Fractional utilization of VO2max measured during a 15-minute performance test
Hemoglobin mass | Changes from before the intervention to immediately after the intervention
  Hemoglobin mass measured using CO rebreathing (g)
Blood volume | Changes from before the intervention to immediately after the intervention
  Blood volume measured using CO rebreathing
Plasma volume | Changes from before the intervention to immediately after the intervention
  Plasma volume measured using CO rebreathing
Red blood cell volume | Changes from before the intervention to immediately after the intervention
  Red blood cell volume measured using CO rebreathing
Hematocrit | Changes from before the intervention to immediately after the intervention
  Hematocrit measured using centrifugation

OTHER OUTCOMES:
Endurance training volume | Throughout study completion (daily), an average of ten weeks
  Self-reported endurance training volume measured as time-spent in different exercise intensity zones
Resistance training volume | Throughout study completion (daily), an average of ten weeks
  Self-reported resistance training volume measured as load x repetitions

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Lofthus, Study Chair — Research Administrator
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Inland Norway, Norway